CLINICAL TRIAL: NCT03022877
Title: Acute and Chronic Protective Effects of Peri-interventional Administration of Levosimendan in ST Elevation Myocardial Infarctions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Rationale obsolete
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Levo-STEMI
Record Dates: First submitted 2017-01-06; First posted 2017-01-18 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Myocardial Infarction; Outcome
MeSH Terms: conditions — Myocardial Infarction | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo is given as a Bolus (instead of Bolus application of Levosimendan) over 10 min i.v., starting 10 min before recanalization.
  Interventions: Drug: Levosimendan
- Bolus Levosimendan (Active Comparator): Levosimendan is given as Bolus (12 µg/kg over 10 min i.v.), starting 10 min before recanalization.
  Interventions: Drug: Levosimendan
- Bolus and infusion Levosimendan (Active Comparator): Levosimendan is given as Bolus (12 µg/kg over 10 min i.v.), starting 10 min before recanalization and additionally as continuous infusion (0.1-0.2 µg/kg/min i. v. for 24 hours).
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — In a prospective randomized setting, patients are included with an acute STEMI of the anterior wall. A bolus administration Levosimendan with/without following continuous infusion over 24 hours compared to a control group (placebo) will be examined. The initiation of therapy is carried out for 10 min. prior to reperfusion. The coronary Intervention is performed immediately after inclusion at the latest within 6 hours after the onset of symptoms. The administration of Levosimendan is based on a fixed schema: Bolus: 12 µg/kg over 10 min I. V., starting 10 min before recanalization and an addition of 0.1-0.2 µg/kg/min i. v. for 24 hours in the continuous infusion group.

SUMMARY:
In the proposed project the investigators want to assess whether the approach of the post-conditioning by Levosimendan in patients with acute STEMI is safe and reproducible, can be used with a positive influence on the outcomes with respect to myocardial damage, cardiac left ventricular remodeling, myocardial function, the occurrence of cardiac events and quality of life.

DETAILED DESCRIPTION:
An acute ST-elevation myocardial infarction (STEMI) is a severe disease that triggers an adverse remodeling, and served in progressive heart failure with a case fatality rate of 50% in 5 years. The opening of the occluded vessel is the first and most important therapy, the reperfusion improved both the function as well as the long-term survival. At the same time, experimental and clinical studies show, however, that this reperfusion self-reinforced damage of the myocardium. An additional Intervention in this trigger phase could not only reduce the acute damage, but long-term protective effects. Both effects could be an approach for the Calcium-Sensitizer Levosimendan in the animal model. So far, no clear effect on the remodeling and survive was demonstrated after myocardial infarction in the clinic. This could be mainly due to the delayed application in relation to the reperfusion and on the selection of suitable methods for the presentation of the effects on myocardial structure and function. In the proposed project the investigators want to assess whether the approach of the post-conditioning by Levosimendan in patients with acute STEMI is safe and reproducible, can be used with a positive influence on the outcomes with respect to myocardial damage, cardiac left ventricular remodeling, myocardial function, the occurrence of cardiac events and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* STEMI of the anterior wall < 6 hrs
* capacity to Consent

Exclusion Criteria:

* previous myocardial infarction or bypass surgery
* relevant vitium
* STEMI of the posterior wall
* any contraindications to MRI
* unstable hemodynamics (hypotension, catecholamine therapy, severe arrhythmia), -respiratory failure
* onset of symptoms more than 6 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of the increase in left ventricular end-diastolic volume index (LVEDVi) | 12 months after coronary intervention due to the infarction
  echocardiography and MRI examinations (LVEDVi) and comparison between baseline and 12 months data

SECONDARY OUTCOMES:
Size of the acute myocardial damage due to the infarction | 12 months after coronary intervention due to the infarction
  MRI examination (infarction area) and comparison between baseline and 12 months data
Event-free survival | 12 months after coronary intervention due to the infarction
  collection of data from the patient after 12 months about adverse events as myocardial infarction, stroke, revascularization and death
functional changes (imaging) | 12 months after coronary intervention due to the infarction
  echocardiography and MRI examinations about LV function
structural changes | 12 months after coronary intervention due to the infarction
  MRI examinations about fibrosis
functional changes (spirometry) | 12 months after coronary intervention due to the infarction
  changes of capacity by spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, Principal Investigator — Cardiology, RWTH University Hospital Aachen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks GC, Lee BK, Rao R, Lin F, Morin DP, Zweibel SL, Buxton AE, Pletcher MJ, Vittinghoff E, Olgin JE; PREDICTS Investigators. Predicting Persistent Left Ventricular Dysfunction Following Myocardial Infarction: The PREDICTS Study. J Am Coll Cardiol. 2016 Mar 15;67(10):1186-1196. doi: 10.1016/j.jacc.2015.12.042. PMID 26965540
- [Result] Kloner RA, Jennings RB. Consequences of brief ischemia: stunning, preconditioning, and their clinical implications: part 2. Circulation. 2001 Dec 18;104(25):3158-67. doi: 10.1161/hc5001.100039. PMID 11748117
- [Result] Yellon DM, Hausenloy DJ. Myocardial reperfusion injury. N Engl J Med. 2007 Sep 13;357(11):1121-35. doi: 10.1056/NEJMra071667. No abstract available. PMID 17855673
- [Result] du Toit EF, Smith W, Muller C, Strijdom H, Stouthammer B, Woodiwiss AJ, Norton GR, Lochner A. Myocardial susceptibility to ischemic-reperfusion injury in a prediabetic model of dietary-induced obesity. Am J Physiol Heart Circ Physiol. 2008 May;294(5):H2336-43. doi: 10.1152/ajpheart.00481.2007. Epub 2008 Mar 21. PMID 18359896
- [Result] Hein M, Roehl AB, Baumert JH, Scherer K, Steendijk P, Rossaint R. Anti-ischemic effects of inotropic agents in experimental right ventricular infarction. Acta Anaesthesiol Scand. 2009 Aug;53(7):941-8. doi: 10.1111/j.1399-6576.2009.01994.x. Epub 2009 May 6. PMID 19426242
- [Result] Kin H, Zhao ZQ, Sun HY, Wang NP, Corvera JS, Halkos ME, Kerendi F, Guyton RA, Vinten-Johansen J. Postconditioning attenuates myocardial ischemia-reperfusion injury by inhibiting events in the early minutes of reperfusion. Cardiovasc Res. 2004 Apr 1;62(1):74-85. doi: 10.1016/j.cardiores.2004.01.006. PMID 15023554
- [Result] Qarawani D, Cohen A, Nahir M, Hasin Y. Facilitation of left ventricular function recovery post percutaneous coronary intervention by levosimendan. Int J Cardiol. 2013 Sep 20;168(1):237-42. doi: 10.1016/j.ijcard.2012.09.088. Epub 2012 Oct 11. PMID 23063476